CLINICAL TRIAL: NCT05173168
Title: A Pilot Study to Assess the Safety Profile of resB®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResBiotic Nutrition, Inc. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESB101
Record Dates: First submitted 2021-11-16; First posted 2021-12-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Healthy; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic Dietary Supplement (Experimental): resB® Lung Support - 1 capsule 2x daily for 4 weeks
  Interventions: Dietary Supplement: Probiotic Dietary Supplement

INTERVENTIONS:
Dietary Supplement: Probiotic Dietary Supplement — Probiotic dietary supplement containing 3 probiotic strains and 3 herbal extracts
  Other Names: resB® Lung Support

SUMMARY:
The study investigates the safety and tolerability of 4-week, twice daily supplementation of resB® Lung Support in asthma patients and healthy participants.

DETAILED DESCRIPTION:
resB® Lung Support is a probiotic dietary supplement that contains 3 probiotic strains and 3 herbal extracts: turmeric, holy basil, and vasaka. The proprietary herbal and probiotic blend is formulated to support proper lung structure and function. The study investigates the safety and tolerability of twice-daily supplementation of resB® Lung Support in asthma patients and healthy participants for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be between 18 - 65 years.
3. Has a stable body weight (≤5 % change) over the past 3-months.
4. Is in general good health, as determined by the investigator.
5. Avoid consuming probiotics within 12 weeks prior to baseline visit, until the end of the trial.
6. Has asthma and on stable medication for at least 3 months (confirmed by prescribed medication) AND/OR be general good health at the discretion of the investigator.
7. Maintain current level of physical activity.
8. Willing to consume the investigational product daily for the duration of the trial.

Exclusion Criteria:

1. Are less than 18 or greater than 65.
2. Participants who are pregnant, breastfeeding, or wish to become pregnant during the trial.
3. Participants currently of child-bearing potential, but not using an effective method of contraception, as outlined below:

   1. Complete abstinence from intercourse two weeks prior to administration of the investigational product, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the investigational product in cases where participant discontinues the trial prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
   2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that participant.
   3. Sexual partner(s) is/are exclusively female.
   4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g. male condom, female diaphragm) or contraceptive pill. The participant must be using this method for at least 1 week following the end of the trial.
   5. Use of any non-hormonal intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1 % per year. The participant must have the device inserted at least 2 weeks prior to the first Screening Visit, throughout the trial, and 2 weeks following the end of the trial.
4. Are hypersensitive or known allergy to any of the components of the investigational product.
5. Has taken antibiotics within the previous 12 weeks.
6. Has taken probiotics within the previous 12 weeks.
7. Has taken oral steroids (>10 mg/day) for more than 3 days in the previous 12 weeks.
8. Taking any immunosuppressive medications which in the opinion of the investigator are likely to have an impact on the outcomes of the trial.
9. Has made any major dietary changes in the 30 days prior to enrolment.
10. Change in medications or supplements in the 30 days prior to enrolment.
11. Have an acute or chronic illness (e.g., heart disease, inflammatory bowel disease, cancer, HIV) that, in the Investigators judgment, precludes involvement in the study
12. No more than 2 hospital admissions in the previous 6 months asthma population)
13. Presence of the following in a urine drug screen- Amphetamine/Ecstasy; Benzodiazepines; 6-Monoacetyl Morphine (6-MAM); Cocaine; Creatinine; EDDP; Opiates; Tricyclic Antidepressants; pH Detect
14. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
15. Participants may not be receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than 3-months prior to this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing at least one adverse event (AE) | 0-4 weeks
Number of AEs including causality, severity, and seriousness assessments | 0-4 weeks
Number of participants with discontinuations due to AEs | 0-4 weeks
Number of participants with clinically significant changes in vital signs as a measure of safety | Baseline, Week 2, Week 4
  Number of participants with clinically significant changes in vital signs including systolic blood pressure (mmHg), diastolic blood pressure (mmHg), heart rate (BPM), and body temperature will be reported.
Number of participants with clinical laboratory abnormalities as a measure of safety | Baseline, Week 2, Week 4
  Number of participants with clinical laboratory abnormalities (clinical laboratory tests include the following: hematology panel, serum chemistry panel) will be reported.

OTHER OUTCOMES:
St George's Respiratory Questionnaire (SGRQ) | 0-4 weeks
  Change in SGRQ total score
Gut microbiota | 0-4 weeks
  Change in gut microbiota (16s sequencing)
Serum MMP-9 | 0-4 weeks
  Change in serum Matrix Metallopeptidase-9 (MMP-9)
Cytokines (IL-1ß, IL-6, IL-8 & TNF-α) | 0-4 weeks
  Change in inflammatory cytokines (IL-1ß, IL-6, IL-8 & TNF-α)
Serum Vitamin D | 0-4 weeks
  Change in serum vitamin D (ng/mL)
Lung function | 0-4 weeks
  Change in lung function measured by spirometry (Forced Expired Volume in 1 second [FEV2]/Forced Vital Capacity [FVC])
Oxygen levels | 0-4 weeks
  Change in oxygen levels (% percentage pulse oxygen levels)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Clinical Trials, 1st Floor, Block C, Heron House, Retail Park, Blackpool, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wenger NM, Qiao L, Nicola T, Nizami Z, Martin I, Halloran BA, Tanaka K, Evans M, Xu X, Dinan TG, Kakilla C, DunnGalvin G, Ambalavanan N, Willis KA, Gaggar A, Lal CV. Clinical trial of a probiotic and herbal supplement for lung health. Front Nutr. 2023 Jun 13;10:1168582. doi: 10.3389/fnut.2023.1168582. eCollection 2023. PMID 37384109